CLINICAL TRIAL: NCT06468020
Title: The Effect of the Gather.Town Gaming Intervention for Promoting Depression Literacy Among Pregnant Adolescents in Thailand
Brief Title: Gather.Town Gaming for Pregnant Adolescents With Depression Literacy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University (Other)
Responsible Party: Principal Investigator, Chotip Phonkusol, Principal Investigator, National Taiwan University
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: The Gather.town gaming
Record Dates: First submitted 2024-05-07; First posted 2024-06-21 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Gamification
Keywords: Pregnant adolescents; Depression literacy; Game-based learning; Gather.town; Digital mental health intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Gather.town gaming intervention (Experimental): The Gather.town intervention, based on Rational Emotive Behavior Therapy (REBT), was delivered over four weeks with two 40-50-minute sessions per week, totaling eight sessions. Conducted via laptops or desktops at antenatal care clinics, the program began with baseline assessments and distribution of a booklet. Participants were introduced to the Gather.town platform. Each session included a homework review (except Sessions 1 and 8), a brief educational video (excluding Session 2), and an interactive game guided by the avatar "Sati." Session 2 focused on scenario analysis to link thoughts, emotions, and behaviors. All sessions ended with debriefing, homework, and written reflection. Sessions 5 and 6 featured virtual relaxation practices. The final session included post-assessments and a closing activity. Participants also received routine antenatal care throughout.
  Interventions: Other: The Gather.town gaming intervention
- Control group (No Intervention): Participants in the control group will receive a booklet and routine care that is regularly available in the health system for both adult and adolescent pregnant women. Antenatal care is provided by nurses in the antenatal care unit and includes health assessments and educational classes covering topics such as nutrition, exercise, sexual intercourse, fetal movement monitoring, childbirth preparation, and breastfeeding. Participants are expected to attend at least five antenatal visits throughout their pregnancy: the first visit should occur before 12 weeks of gestation, with subsequent visits at 18, 26, 32, and 38 weeks.

INTERVENTIONS:
Other: The Gather.town gaming intervention — The online game-based learning intervention (oGBL): The investigator will develop the oGBL intervention based on Rational Emotive Behavior Therapy (REBT), which consists of 8 sessions and plays a game through the Gather.Town platform.
  Arms: The Gather.town gaming intervention

SUMMARY:
Aim

The study seeks to:

1. To assess the effect of the Gather.town gaming intervention on promoting depression literacy among pregnant adolescents in Thailand.
2. To compare the depression literacy before and after receiving the Gather.town gaming intervention in the experimental group.

Methods This quasi-experimental study employed a two-group, pretest-posttest design to assess the effect of a Gather.town gaming intervention on promoting depression literacy among pregnant adolescents in Thailand. 64 first-time pregnant adolescents aged 15-19 years with gestational age under 21 weeks were recruited from three hospitals using stratified random sampling. Participants were randomly assigned to the experimental group (n = 32) or control group (n = 32).

The experimental group participated in eight sessions of REBT-based interactive gaming on the Gather.town platform over four weeks (two sessions per week), while the control group received routine antenatal care and a depression literacy booklet. Quantitative data were collected at four time points (baseline, immediate post-intervention, 1-month, and 3-month follow-ups) using validated tools, including the Depression Literacy Questionnaire (D-Lit), depressive symptoms (EPDS), mental distress (BSRS-5), and platform usability (SUS). Qualitative data were gathered through focus group interviews after the intervention. Statistical analyses were performed using SPSS version 22. Descriptive statistics summarized participant characteristics. Chi-square tests examined group differences. Generalized Estimating Equations (GEE) were used to compare depression literacy scores across time points while accounting for clustering by hospital and adjusting for covariates. The significance level was set at p < 0.05.

DETAILED DESCRIPTION:
Measurement

1. The researcher has developed this information based on a review of the literature, consisting of 17 questions. These include six items on socio-demographic information: age, educational level, marital status, current living situation, employment status, and household monthly income. There are 11 items related to health information, including week of pregnancy, pregnancy planning, history of abortion, number of abortions, abnormal symptoms during pregnancy, history of alcohol drinking, history of cigarette/e-cigarette smoke, stress coping behaviors, help-seeking behavior for emotional problems, sources of mental health support, and sources of payment for health care.
2. The Depression Literacy Questionnaire (D-Lit) will be used to evaluate an individual's level of depression literacy, covering incidence, recognition of depressive symptoms, differentiation of symptoms from other mental illnesses, non-medication effectiveness, and knowledge of medication. The questionnaire consists of 22 true-or-false items. Respondents can answer each item with one of three options: "true," "false," or "don't know." Each correct response receives one point, while "don't know" is counted as an incorrect response. In this study, one question from the original version-"Not stepping on cracks in the footpath may be a sign of depression"-was omitted as it was not culturally suitable for the Thai context. The overall score ranges from 0 to 21, with higher scores representing higher depression literacy levels. The scale has a Cronbach's alpha coefficient of 0.70.
3. The Edinburgh Postnatal Depression Scale (EPDS) was designed to screen for depressive symptoms among postpartum women in a community setting. Meanwhile, the EPDS is also a widely accepted instrument for screening depression in the prenatal period. This scale consists of 10 items to assess depressive symptoms, including mood changes, anxiety, and self-harm ideation, over the past 7 days. Respondents are asked to rate how often they experienced each symptom in the past week on a 4-point Likert scale, with scores of 0, 1, 2, and 3 assigned based on the severity of the symptoms. Items 3 and 5 to 10 are reverse-scored (3, 2, 1, and 0). The total score is calculated by summing each of the ten items, with possible scores ranging from 0 to 30. A cut-off score of 12 or 13 indicates those likely to be suffering from depression. Psychometrically, the EPDS scale demonstrates good construct validity and high internal consistency reliability in primary care and clinical settings, with Cronbach's alpha values of 0.87. The cut-off score of the Thai version of the EPDS is suitable for diagnosing depression among pregnant women at ≥ 11, with an acceptable Cronbach's alpha of 0.77.
4. The 5-item Brief Symptom Rating Scale (BSRS-5) is commonly used for screening psychological disorders. It consists of 5 self-rated items measuring brief psychological symptoms, including insomnia, anxiety, hostility, depression, and inferiority. Each item is rated on a Likert scale ranging from 0 (not at all) to 4 (extremely). A total score on the BSRS-5 of more than 15 indicates severe mental distress; scores between 10 and 14 indicate moderate distress, scores between 6 and 9 indicate mild distress, and scores lower than 6 indicate normal status. The scale has a Cronbach's alpha coefficient ranging from 0.77 to 0.90. In this sub-study, the researcher will translate the scale into Thai and have it back-translated by two experts proficient in both English and Thai.
5. The System Usability Scale (SUS) will be used to measure the usability of the Gather.town platform. The scale of SUS consists of 10 simple questions. The respondents are asked to rate how they perceive usability on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The total score ranges with the range of possible scores from 0 to 100. A score less than 51 indicates system usability at a minimum level, 51-68 points mean system usability at a low level, 68 points represent a moderate level of system usability, 68-80.3 points suggest system usability at a good level, and scores more than 80.3 points represent an excellent level of system usability. The SUS has demonstrated good construct validity and high reliability, with an acceptable Cronbach's alpha from 0.77 to 0.97.
6. Pre-intervention survey We will ask three open-ended questions before the intervention: "Have you heard of the Gather.town platform before?", "What are your expectations for the Gather.town gaming intervention for mental health support during pregnancy?", and "What features or activities would you like in the Gather.town gaming intervention to help you cope with stress during pregnancy?". These questions aim to gather pregnant adolescents' opinions and expectations for addressing mental health problems via the Gather.town gaming intervention.
7. Qualitative feedback collected after each session of the program After each session of the program, we will add three open-ended questions to obtain qualitative initial feedback from pregnant adolescents: "What did you like the most about the Gather.town gaming intervention?", "What did you not like about the Gather.town gaming intervention?", and "What suggestions do you have to improve the Gather.town gaming intervention?"
8. Qualitative reflection collected after the intervention via the focus group interview For the focus group interview after the intervention, we will add three open-ended questions to explore participants' experiences with the Gather.town gaming intervention and its impact on their depression literacy. "How have your knowledge and beliefs about depression changed after participating in the Gather.town gaming intervention?", "What aspects of the Gather.town intervention did you find most helpful in improving your understanding of depression?", and "How has the Gather.town gaming intervention influenced your attitude toward seeking help for mental health?"

ELIGIBILITY:
Inclusion Criteria:

1. First-time pregnant adolescents aged 15-19 years with gestational ages not exceeding 21 weeks.
2. Being able to read Thai and use a computer or laptop to operate the intervention materials.

Exclusion Criteria:

1. Being unwilling to participate in this study.
2. Being unable to adhere to the entire intervention process or follow-up.
3. Self-reported psychiatric diagnosis of any severe mental illnesses, i.e., major depression, schizophrenia, or bipolar disorder.

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the knowledge of depression, as measured by a true or false questionnaire of the Depression Literacy Questionnaire (D-Lit) | Baseline, immediately after the intervention, and at the 1-month and 3-month follow-ups
  Scores are measured using a true or false questionnaire, with one point awarded for each correct answer. The score ranges from 0 to 21, with higher scores indicating greater knowledge.

SECONDARY OUTCOMES:
Change from baseline in mental distress levels, as measured by the Likert scale of the 5-item Brief Symptom Rating Scale (BSRS-5) | Baseline, immediately, and after the intervention
  Scores are measured on a Likert scale ranging from 0 to 4. The total score ranges from 0 to 20, with scores more than 15 indicating severe mental distress, scores between 10 and 14 indicating moderate distress, scores between 6 and 9 indicating mild distress, and scores lower than 6 indicating normal status.
Change from baseline in depression levels, as measured by the Likert scale of The Edinburgh Postnatal Depression Scale (EPDS) | Baseline, immediately, and after the intervention
  Scores are measured on a Likert scale ranging from 0 to 3. The total score ranges from 0 to 30, with ≥ 11 indicating likely to be suffering from depression
To measure the usability of the Gather.town platform, as measured by the Likert scale of the System Usability Scale (SUS) | immediately after the intervention
  Scores are measured on a Likert scale ranging from 1 to 5. The total score ranges from 0 to 100, with higher total scores indicating a good level of system usability

CONTACTS AND LOCATIONS:
Overall Officials: Chotip Phonkusol, Principal Investigator — National Taiwan University

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Starting in June 2025
Access Criteria: The information on the study protocol will be shared with other researchers.